CLINICAL TRIAL: NCT04679090
Title: Do Physical Activity Levels Predict Functional Improvements Following a Structured Exercise Program for Women Living With Breast Cancer?
Brief Title: Physical Activity Levels and Functional Improvement in Breast Cancer Survivors
Acronym: CanEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of New Brunswick (Other)
Collaborators: Ultramar (Unknown); Quebec Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: University Brunswick
Record Dates: First submitted 2020-12-01; First posted 2020-12-22 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant (Experimental): Participants will answer a series of questionnaires, wear a physical activity tracker (pedometer) and do functional tests (six minute walk test, chair stand test, balance, back scratch, sit and reach, leg strength and hand strength) pre and post.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Participants will exercise twice a week for twelve weeks total.

SUMMARY:
The main objective of our project is to describe what characteristics (e.g., age, current physical activity level) women present when starting the exercise program are potentially associated with an improvement in functional abilities measured with different tests such as the distance you can cover while walking for six minutes.

DETAILED DESCRIPTION:
The main research objective is to investigate the relationship between baseline physical activity and improvement in physical function, quantified using changes in 6-minute walk test (6MWT) results over the course of the 12-week program. An association is hypothesized to exist between the two variables even when adjusted for weeks into treatment. The goal of the 6MWT is to cover as much distance as possible in six minutes, using as many breaks s necessary. The test is often performed using a 20-meter hallway but requires no specific equipment. A recent study reported that the result of the 6MWT could be used as a measure of the major components of global health in women with breast cancer, making its use in our research especially relevant. Aside from physical functions, baseline characteristics will also be used to determine what characteristics, if any, are associated with health and psychosocial outcomes such as quality of life, social connectedness/support, and mental well-being. The data collected is certain to fill a gap in the literature, and will therefore be likely published in an important journal in the field.

ELIGIBILITY:
Inclusion Criteria:

* Have received a diagnosis of breast cancer in your lifetime
* 19 years of age and older
* Cleared by medical team to participate in the study
* Have the intention to exercise at the facility for the duration of the study

Exclusion Criteria:

-

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Pre and post (after 12 weeks)
  6-minute walk test (meters walked)
Balance | Pre and post (after 12 weeks)
  One leg stand test (seconds)
Strength, Hand grip | Pre and post (after 12 weeks)
  Amount of force that can be exerted during grip squeeze (kg)
Strength, Chair stand test | Pre and post (after 12 weeks)
  Chair stand test, number of chair stand in 30 seconds
Flexibility, back scratch test | Pre and post (after 12 weeks)
  Back scratch test (cm)
Flexibility, sit and reach | Pre and post (after 12 weeks)
  Sit and reach test
Physical Activity Level | Pre and post (after 12 weeks)
  Pedometer to determine minutes in moderate-vigorous physical activity and steps per day

SECONDARY OUTCOMES:
Attendance | Pre and post (after 12 weeks)
  Amount of exercise sessions attended during the 12-week program
Weight | Pre and post (after 12 weeks)
  Weight of individual (kg)
Height | Pre and post (after 12 weeks)
  Height of individual (cm)
Resting Blood Pressure | Pre and post (after 12 weeks)
  Systolic and diastolic blood pressure (mmHg)
Resting Heart Rate | Pre and post (after 12 weeks)
  Resting heart rate (beats per minute)
Body-mass Index | Pre and post (after 12 weeks)
  Measure of body fat based on height and weight (kg/m^2)
Waist Circumference | Pre and post (after 12 weeks)
  Measurement around the waist (cm)
FANTASTIC Lifestyle Checklist | Pre and post (after 12 weeks)
  Meaningful improvement above day-to-day variability on the 6MWT
Functional Assessment of Cancer Therapy General (FACT - G) | Pre and post (after 12 weeks)
  27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being
Functional Assessment of Cancer Therapy Fatigue (FACT - F) | Pre and post (after 12 weeks)
  40-item measure that assesses self-reported fatigue and its impact upon daily activities and function
Depression Anxiety Stress Scales (DASS) | Pre and post (after 12 weeks)
  42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress.
Pittsburgh Sleep Quality Index (PSQI) | Pre and post (after 12 weeks)
  A self-report questionnaire that assesses sleep quality over a 1-month time interval
Godin-Shephard Leisure-Time Physical Activity Questionnaire | Pre and post (after 12 weeks)
  Questionnaire used to identify self-reported leisure-time physical activity
Age | Pre and post (after 12 weeks)
  Age (years)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Bouchard, Principal Investigator — University of New Brunswick
Locations (3):
- Canada (3):
  - University of New Brunswick, Fredericton, New Brunswick
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - University of Prince Edward Island, Charlottetown, Prince Edward Island